CLINICAL TRIAL: NCT03467958
Title: A Phase 3, Multicenter, Open-Label Extension Study of Oral Ozanimod for Moderately to Severely Active Crohn's Disease
Brief Title: An Extension Study of Oral Ozanimod for Moderately to Severely Active Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC01-3204; U1111-1203-8203 (Registry Identifier: WHO); 2017-004295-55 (EudraCT Number)
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Crohn Disease; Oral; Ozanimod; Moderately active; Severely active; RPC01; RPC01-3204
MeSH Terms: conditions — Crohn Disease | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of oral Ozanimod (Experimental)
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days

SUMMARY:
This is an extension study to evaluate safety and efficacy of ozanimod in participants with moderately to severely active Crohn's Disease.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Is not in clinical response or clinical remission after completing 12 weeks in the Induction Studies
* Experience relapse or who complete the Maintenance Study
* Complete a study of ozanimod for Crohn's Disease and meet the criteria for participation

Exclusion Criteria:

* Has any clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, psychiatric, or other major systemic disease making implementation of the protocol or interpretation of the study difficult or that would put the subject at risk by participating in the study
* Has suspected or diagnosed intra-abdominal or perianal abscess that has not been appropriately treated
* Is receiving treatment with any of the following drugs or interventions: CYP2C8 inducers; Monoamine oxidase inhibitors

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (766):
- United States (190):
  - Holland Center for Family Health, Peoria, Arizona
  - Local Institution - 202, Scottsdale, Arizona
  - Local Institution - 026, North Little Rock, Arkansas
  - Local Institution - 284, Camarillo, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Local Institution - 039, Garden Grove, California
  - Ucsd Medical Center, La Jolla, California
  - San Diego Clinical Trials, La Mesa, California
  - Local Institution - 010, Lancaster, California
  - Local Institution - 061, Los Angeles, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Matrix Clinical Research Inc, Los Angeles, California
  - Local Institution - 110, Los Angeles, California
  - Facey Medical Foundation (Parent), Mission Hills, California
  - ABS Health, LLC, Mission Viejo, California
  - Alliance Clinical Research, Oceanside, California
  - Local Institution - 027, Orange, California
  - Palo Alto Center-Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Havana Research Institute LLC, Pasadena, California
  - Local Institution - 006, Rialto, California
  - Sutter Medical Group, Roseville, California
  - Local Institution - 280, Sacramento, California
  - Local Institution - 003, San Diego, California
  - Local Institution - 281, San Francisco, California
  - New Hope Research Development, West Covina, California
  - Local Institution - 065, Colorado Springs, Colorado
  - Local Institution - 297, Lakewood, Colorado
  - Local Institution - 182, Bristol, Connecticut
  - Local Institution - 225, Bristol, Connecticut
  - Local Institution - 091, New Haven, Connecticut
  - Local Institution - 062, Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - South Lake Pain Institute, Clermont, Florida
  - American Research Institute Inc, Cutler Bay, Florida
  - Local Institution - 112, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Local Institution - 218, Gainesville, Florida
  - Local Institution - 203, Hialeah, Florida
  - Floridian Clinical Research LLC, Hialeah, Florida
  - Harmony Medical Research Institute, Hialeah, Florida
  - Local Institution - 179, Hollywood, Florida
  - Vista Health Research, Homestead, Florida
  - SIH Research, Kissimmee, Florida
  - Local Institution - 016, Largo, Florida
  - Local Institution - 067, Lighthouse PT, Florida
  - Center For Advanced Gastroenterology, Maitland, Florida
  - LMG Research, Miami, Florida
  - Local Institution - 199, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Local Institution - 169, Miami, Florida
  - Local Institution - 175, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Local Institution - 044, Miami Springs, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Local Institution - 192, New Port Richey, Florida
  - Local Institution - 214, New Smyrna Beach, Florida
  - Local Institution - 200, Orlando, Florida
  - Local Institution - 076, Orlando, Florida
  - Local Institution - 002, Palmetto Bay, Florida
  - Theia Clinical Research, LLC, Pinellas Park, Florida
  - Local Institution - 098, Port Orange, Florida
  - Precision Clinical Research, LLC., Sunrise, Florida
  - Local Institution - 183, Tampa, Florida
  - Apex Clinical Research, Tampa, Florida
  - Local Institution - 226, Tampa, Florida
  - Local Institution - 107, Tampa, Florida
  - Local Institution - 149, Tampa, Florida
  - Local Institution - 114, Weeki Wachee, Florida
  - Consultative Gastroenterology, Atlanta, Georgia
  - Local Institution - 037, Atlanta, Georgia
  - Local Institution - 220, Atlanta, Georgia
  - Local Institution - 222, Atlanta, Georgia
  - Local Institution - 019, Atlanta, Georgia
  - Local Institution - 063, Atlanta, Georgia
  - Local Institution - 074, Columbus, Georgia
  - Local Institution - 143, Decatur, Georgia
  - Local Institution - 028, Macon, Georgia
  - Local Institution - 115, Idaho Falls, Idaho
  - Local Institution - 194, Chicago, Illinois
  - Local Institution - 036, Chicago, Illinois
  - Local Institution - 022, Chicago, Illinois
  - Local Institution - 216, Oak Lawn, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Local Institution - 092, Evansville, Indiana
  - Local Institution - 033, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Local Institution - 070, Topeka, Kansas
  - Local Institution - 155, Lexington, Kentucky
  - Local Institution - 020, Baton Rouge, Louisiana
  - CroNOLA LLC, Houma, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Clinical Trials of SW Louisiana LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Nola Research Works, New Orleans, Louisiana
  - Local Institution - 278, Baltimore, Maryland
  - Local Institution - 129, Catonsville, Maryland
  - Local Institution - 282, Glen Burnie, Maryland
  - Local Institution - 142, Chestnut Hill, Massachusetts
  - Local Institution - 228, North Worcester, Massachusetts
  - Local Institution - 286, Springfield, Massachusetts
  - Local Institution - 024, Worcester, Massachusetts
  - Local Institution - 191, Caro, Michigan
  - Local Institution - 167, Kalamazoo, Michigan
  - Local Institution - 005, Novi, Michigan
  - Local Institution - 108, Southfield, Michigan
  - Local Institution - 301, Wyoming, Michigan
  - Local Institution - 300, Ypsilanti, Michigan
  - Local Institution - 095, Minneapolis, Minnesota
  - Local Institution - 045, Rochester, Minnesota
  - Local Institution - 274, Jackson, Mississippi
  - Local Institution - 198, Kansas City, Missouri
  - Local Institution - 029, St Louis, Missouri
  - Internal Medicine Specialists, Las Vegas, Nevada
  - Local Institution - 040, Lebanon, New Hampshire
  - Local Institution - 215, Englewood, New Jersey
  - Local Institution - 144, Brooklyn, New York
  - Local Institution - 009, Great Neck, New York
  - Local Institution - 054, Hartsdale, New York
  - Weill Cornell Medical College, New York, New York
  - Concorde Medical Group, New York, New York
  - Local Institution - 105, New York, New York
  - TrialSpark, New York, New York
  - Local Institution - 043, New York, New York
  - Local Institution - 060, North Massapequa, New York
  - Circuit Clinical, Orchard Park, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Local Institution - 017, Asheville, North Carolina
  - Local Institution - 152, Charlotte, North Carolina
  - Local Institution - 055, Charlotte, North Carolina
  - Local Institution - 156, Charlotte, North Carolina
  - Local Institution - 133, Greenville, North Carolina
  - Local Institution - 302, Raleigh, North Carolina
  - Local Institution - 052, Winston-Salem, North Carolina
  - Great Lakes Medical Research, LLC, Beachwood, Ohio
  - Local Institution - 291, Cincinnati, Ohio
  - Local Institution - 018, Cleveland, Ohio
  - Local Institution - 170, Dayton, Ohio
  - Local Institution - 049, Hilliard, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Local Institution - 141, Middleburg Heights, Ohio
  - Great Lakes Medical Research, LLC, Warren, Ohio
  - Local Institution - 087, Norman, Oklahoma
  - Local Institution - 294, Oklahoma City, Oklahoma
  - Local Institution - 208, Oklahoma City, Oklahoma
  - Local Institution - 131, Oklahoma City, Oklahoma
  - Local Institution - 185, Tulsa, Oklahoma
  - Local Institution - 217, Tulsa, Oklahoma
  - Local Institution - 113, Portland, Oregon
  - Local Institution - 197, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Penn State University Milton S Hershey Medical Center, State College, Pennsylvania
  - Local Institution - 253, Providence, Rhode Island
  - Local Institution - 289, Charleston, South Carolina
  - Local Institution - 212, Orangeburg, South Carolina
  - Local Institution - 121, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - Local Institution - 158, Austin, Texas
  - Local Institution - 034, Fort Sam Houston, Texas
  - Local Institution - 056, Houston, Texas
  - Local Institution - 150, Houston, Texas
  - Biopharma Informatic Inc. Research Center, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - GI Specialists of Houston, Houston, Texas
  - Local Institution - 303, Houston, Texas
  - Local Institution - 088, Houston, Texas
  - Local Institution - 196, Houston, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - Accurate Clinical Research Inc, Pasadena, Texas
  - Local Institution - 071, Richardson, Texas
  - Local Institution - 085, San Antonio, Texas
  - Local Institution - 178, San Antonio, Texas
  - Local Institution - 223, San Antonio, Texas
  - Local Institution - 007, Southlake, Texas
  - Local Institution - 181, Temple, Texas
  - Local Institution - 073, Tyler, Texas
  - Local Institution - 292, Riverton, Utah
  - Local Institution - 025, Salt Lake City, Utah
  - Local Institution - 189, Gainesville, Virginia
  - Local Institution - 030, Lynchburg, Virginia
  - Local Institution - 298, Manassas, Virginia
  - Summit Clinical Research, LLC, Petersburg, Virginia
  - The Gastroenterology Group, Reston, Virginia
  - Local Institution - 072, Richmond, Virginia
  - Local Institution - 172, Roanoke, Virginia
  - Virginia Gastroenterology Institute PC, Suffolk, Virginia
  - Local Institution - 296, Williamsburg, Virginia
  - Local Institution - 125, Spokane, Washington
  - Aurora Health Care Aurora Research, Grafton, Wisconsin
  - Local Institution - 089, La Crosse, Wisconsin
- Argentina (11):
  - Local Institution - 501, Buenos Aires
  - Local Institution - 494, Buenos Aires
  - Local Institution - 571, Buenos Aires
  - Local Institution - 500, Buenos Aires
  - Local Institution - 570, Córdoba
  - Local Institution - 495, Córdoba
  - Local Institution - 569, Mar del Plata
  - Local Institution - 496, Rosario
  - Local Institution - 497, Rosario
  - Local Institution - 502, Rosario, Santa Fe
  - Local Institution - 492, San Miguel de Tucumán
- Australia (25):
  - Local Institution - 310, Concord, New South Wales
  - Local Institution - 319, Kingswood, New South Wales
  - Local Institution - 309, Liverpool, New South Wales
  - Local Institution - 318, New Lambton Heights, New South Wales
  - Local Institution - 323, Wollongong, New South Wales
  - Local Institution - 328, Herston, Queensland
  - Local Institution - 313, Maroorchydore, Queensland
  - Local Institution - 321, North Mackay, Queensland
  - Local Institution - 312, South Brisbane, Queensland
  - Local Institution - 311, Woolloongabba, Queensland
  - Local Institution - 308, Adelaide, South Australia
  - Local Institution - 708, Adelaide, South Australia
  - Local Institution - 307, Bedford Park, South Australia
  - Local Institution - 326, Elizabeth Vale, South Australia
  - Local Institution - 320, Woodville South, South Australia
  - Local Institution - 317, Clayton, Victoria
  - Local Institution - 305, Fitzroy, Victoria
  - Local Institution - 329, Geelong, Victoria
  - Local Institution - 327, Melbourne, Victoria
  - Local Institution - 709, Melbourne, Victoria
  - Local Institution - 316, Murdoch, Western Australia
  - Local Institution - 315, Subiaco, Western Australia
  - Local Institution - 325, Bankstown
  - Local Institution - 330, Box Hill
  - Local Institution - 324, Sydney, NSW
- Austria (4):
  - Local Institution - 726, Innsbruck
  - Local Institution - 727, Sankt Pölten
  - Local Institution - 336, Vienna
  - Local Institution - 725, Vienna
- Belarus (2):
  - Local Institution - 745, Grodno
  - Local Institution - 737, Vitebsk
- Belgium (8):
  - Local Institution - 943, Brasschaat, Antwerpen
  - Local Institution - 940, Brussels
  - Local Institution - 939, Edegem
  - Local Institution - 937, Ghent
  - Local Institution - 942, Leuven
  - Local Institution - 936, Liège
  - Local Institution - 938, Seraing
  - Local Institution - 941, Tournai
- Bosnia and Herzegovina (4):
  - Local Institution - 743, Banja Luka
  - Local Institution - 741, Mostar
  - Local Institution - 738, Sarajevo
  - Local Institution - 742, Sarajevo
- Bulgaria (13):
  - Local Institution - 456, Blagoevgrad
  - Local Institution - 746, Plovdiv
  - Local Institution - 753, Rousse
  - Local Institution - 747, Sofia
  - Local Institution - 750, Sofia
  - Local Institution - 755, Sofia
  - Local Institution - 756, Sofia
  - Local Institution - 752, Sofia
  - Local Institution - 749, Sofia
  - Local Institution - 554, Sofia
  - Local Institution - 748, Sofia
  - Local Institution - 553, Stara Zagora
  - Local Institution - 754, Varna
- Canada (18):
  - Local Institution - 273, Calgary, Alberta
  - Local Institution - 227, Edmonton, Alberta
  - Local Institution - 269, Edmonton, Alberta
  - Local Institution - 263, Kelowna, British Columbia
  - Local Institution - 262, New Westminster, British Columbia
  - Local Institution - 255, Vancouver, British Columbia
  - Local Institution - 267, Vancouver, British Columbia
  - Local Institution - 256, Brandon, Manitoba
  - Local Institution - 261, Winnipeg, Manitoba
  - Local Institution - 268, Bridgewater, Nova Scotia
  - Local Institution - 266, Greater Sudbury, Ontario
  - Local Institution - 252, London, Ontario
  - Local Institution - 251, London, Ontario
  - Local Institution - 264, Toronto, Ontario
  - Local Institution - 257, Toronto, Ontario
  - Local Institution - 271, Vaughan, Ontario
  - Local Institution - 254, Montreal, Quebec
  - Local Institution - 270, Ottawa, Quebec
- Chile (5):
  - Local Institution - 389, Concepción
  - Local Institution - 392, Santiago
  - Local Institution - 387, Santiago
  - Local Institution - 391, Santiago
  - Local Institution - 390, Santiago
- China (36):
  - Local Institution - 423, Changzhou, Jiangsu
  - Local Institution - 369, Shanghai, Shanghai Municipality
  - Local Institution - 419, Chengdu, Sichuan
  - Local Institution - 482, Beijing
  - Local Institution - 467, Beijing
  - Local Institution - 379, Bengbu
  - Local Institution - 485, Changchun
  - Local Institution - 376, Changchun
  - Local Institution - 421, Changsha
  - Local Institution - 378, Changsha
  - Local Institution - 414, Changzhou
  - Local Institution - 422, Fuzhou
  - Local Institution - 478, Guangzhou
  - Local Institution - 472, Guangzhou
  - Local Institution - 486, Guangzhou
  - Local Institution - 470, Hangzhou, Zhejiang
  - Local Institution - 491, Hefei
  - Local Institution - 374, Kunming
  - Local Institution - 383, Luzhou
  - Local Institution - 488, Nanchang
  - Local Institution - 418, Nanjing
  - Local Institution - 375, Nanjing
  - Local Institution - 487, Nanjing
  - Local Institution - 473, Shanghai
  - Local Institution - 380, Shanghai
  - Local Institution - 416, Shanghai
  - Local Institution - 377, Shanghai
  - Local Institution - 458, Taichung City
  - Local Institution - 373, Tianjin
  - Local Institution - 475, Wuhan
  - Local Institution - 474, Wuhan
  - Local Institution - 483, Wuhan
  - Local Institution - 381, Wuxi
  - Local Institution - 415, Xi'an
  - Local Institution - 420, Xi'an
  - Local Institution - 370, Zhengzhou
- Colombia (5):
  - Local Institution - 397, Armenia, Quindío Department
  - Local Institution - 398, Barranquilla
  - Local Institution - 395, Bogotá
  - Local Institution - 396, Cali
  - Local Institution - 394, Medellín
- Croatia (6):
  - Local Institution - 453, Koprivnica
  - Local Institution - 763, Osijek
  - Local Institution - 765, Split
  - Local Institution - 452, Zagreb
  - Local Institution - 762, Zagreb
  - Local Institution - 766, Zagreb
- Czechia (12):
  - Local Institution - 767, Brno
  - Local Institution - 772, Brno
  - Local Institution - 773, Hradec Králové
  - Local Institution - 775, Most
  - Local Institution - 771, Olomouc
  - Local Institution - 774, Pardubice
  - Local Institution - 769, Pilsen
  - Local Institution - 573, Prague
  - Local Institution - 368, Prague
  - Local Institution - 776, Prague
  - Local Institution - 768, Prague
  - Local Institution - 770, Prague
- Denmark (3):
  - Local Institution - 611, Copenhagen
  - Local Institution - 610, Holbæk
  - Local Institution - 609, Nykøbing Falster
- Finland (2):
  - Local Institution - 613, Helsinki
  - Local Institution - 614, Turku
- France (18):
  - Local Institution - 647, Neuilly-sur-Seine, Cedex
  - Local Institution - 638, Amiens
  - Local Institution - 639, Béziers
  - Local Institution - 635, Blois
  - Local Institution - 634, Caen
  - Local Institution - 644, Colombes
  - Local Institution - 711, Créteil
  - Local Institution - 616, Dijon
  - Local Institution - 615, Grenoble
  - Local Institution - 633, Lillie Cedex
  - Local Institution - 646, Marseille
  - Local Institution - 507, Montpellier
  - Local Institution - 632, Nantes
  - Local Institution - 630, Pierre-Bénite
  - Local Institution - 641, Rennes
  - Local Institution - 612, Rouen
  - Local Institution - 631, Saint-Priest-en-Jarez
  - Local Institution - 643, Toulouse
- Georgia (18):
  - Local Institution - 786, Batumi
  - Local Institution - 779, Kutaisi
  - Local Institution - 248, Tbilisi
  - Local Institution - 454, Tbilisi
  - Local Institution - 783, Tbilisi
  - Local Institution - 247, Tbilisi
  - Local Institution - 778, Tbilisi
  - Local Institution - 782, Tbilisi
  - Local Institution - 552, Tbilisi
  - Local Institution - 781, Tbilisi
  - Local Institution - 793, Tbilisi
  - Local Institution - 740, Tbilisi
  - Local Institution - 784, Tbilisi
  - Local Institution - 785, Tbilisi
  - Local Institution - 335, Tbilisi
  - Local Institution - 249, Tbilisi
  - Local Institution - 455, Tbilisi
  - Local Institution - 780, Telavi
- Germany (30):
  - Local Institution - 626, Berlin
  - Local Institution - 629, Berlin
  - Local Institution - 665, Berlin
  - Local Institution - 653, Berlin
  - Local Institution - 648, Berlin
  - Local Institution - 650, Berlin
  - Local Institution - 628, Berlin
  - Local Institution - 664, Brandenburg
  - Local Institution - 732, Dachau
  - Local Institution - 662, Frankfurt
  - Local Institution - 654, Frankfurt
  - Local Institution - 574, Frankfurt am Main
  - Local Institution - 657, Frankfurt am Main
  - Local Institution - 658, Halle
  - Local Institution - 656, Halle
  - Local Institution - 659, Hamburg
  - Local Institution - 652, Hamburg
  - Local Institution - 591, Hanover
  - Local Institution - 649, Keil
  - Local Institution - 337, Leipzig
  - Local Institution - 651, Leipzig
  - Local Institution - 655, Ludwigshafen am Rhein
  - Local Institution - 730, Ludwigshafen am Rhein
  - Local Institution - 660, Mainz
  - Local Institution - 667, Münster
  - Local Institution - 620, Neuruppin
  - Local Institution - 584, Nürtingen
  - Local Institution - 661, Stuttgart
  - Local Institution - 666, Tübingen
  - Local Institution - 663, Ulm
- Greece (8):
  - Local Institution - 790, Athens
  - Local Institution - 588, Athens
  - Local Institution - 791, Athens
  - Local Institution - 792, Athens
  - Local Institution - 592, Athens, Attiki
  - Local Institution - 787, Heraklion
  - Local Institution - 789, Thessaloniki
  - Local Institution - 788, Thessaloniki
- Hong Kong (2):
  - Local Institution - 404, Hong Kong
  - Local Institution - 405, Kowloon
- Hungary (11):
  - Local Institution - 798, Békéscsaba
  - Local Institution - 803, Budapest
  - Local Institution - 804, Budapest
  - Local Institution - 556, Budapest
  - Local Institution - 801, Győr
  - Local Institution - 555, Gyula
  - Local Institution - 797, Miskolc
  - Local Institution - 800, Nagykanizsa
  - Local Institution - 816, Szekszárd
  - Local Institution - 805, Szentes
  - Local Institution - 799, Székesfehérvár
- India (11):
  - Local Institution - 444, Hyderabad, Andhra Pradesh
  - Local Institution - 407, Surat, Gujarat
  - Local Institution - 332, Gurgaon, Haryana
  - Local Institution - 445, Kochi, Kerala
  - Local Institution - 446, Ludhiana, Punjab
  - Local Institution - 443, Jaipur, Rajasthan
  - Local Institution - 399, Jaipur, Rajasthan
  - Local Institution - 408, Coimbatore, Tamil Nadu
  - Local Institution - 331, Hyderabad, Telangana
  - Local Institution - 457, Delhi
  - Local Institution - 411, New Delhi
- Ireland (2):
  - Local Institution - 975, Dublin, Dublin
  - Local Institution - 973, Dublin
- Israel (12):
  - Local Institution - 343, Afula
  - Local Institution - 345, Bat Yam
  - Local Institution - 346, Beer Jacob
  - Local Institution - 350, Haifa
  - Local Institution - 339, Jerusalem
  - Local Institution - 347, Jerusalem
  - Local Institution - 349, Kfar Saba
  - Local Institution - 344, Nahariya
  - Local Institution - 341, Petah Tikva
  - Local Institution - 342, Ramat Gan
  - Local Institution - 338, Rehovot
  - Local Institution - 340, Tel Aviv
- Italy (20):
  - Local Institution - 677, Bologna
  - Local Institution - 684, Brescia
  - Local Institution - 688, Brescia
  - Local Institution - 689, Castellana Grotte
  - Local Institution - 679, Catanzaro
  - Local Institution - 687, Chieti
  - Local Institution - 674, Messina
  - Local Institution - 672, Milan
  - Local Institution - 686, Milan
  - Local Institution - 334, Milan
  - Local Institution - 678, Monza
  - Local Institution - 685, Padua
  - Local Institution - 682, Palermo
  - Local Institution - 673, Pavia
  - Local Institution - 681, Roma
  - Local Institution - 675, Roma
  - Local Institution - 671, Rome
  - Local Institution - 680, Udine
  - Local Institution - 670, Varese
  - Local Institution - 676, Verona
- Latvia (3):
  - Local Institution - 602, Riga
  - Local Institution - 601, Riga
  - Local Institution - 600, Riga
- Lithuania (5):
  - Local Institution - 605, Kaunas
  - Local Institution - 603, Klaipėda
  - Local Institution - 607, Vilnius
  - Local Institution - 606, Vilnius
  - Local Institution - 604, Vilnius
- Mexico (10):
  - Local Institution - 526, Zapapan, Jalisco
  - Local Institution - 532, Monterrey, Nuevo León
  - Local Institution - 525, Monterrey, Nuevo León
  - Local Institution - 447, Monterrey, Nuevo León
  - Local Institution - 449, Monterrey, Nuevo León
  - Local Institution - 529, Querétaro City, Querétaro
  - Local Institution - 528, Chihuahua City
  - Local Institution - 448, Mexico City
  - Local Institution - 527, México
  - Local Institution - 530, Tlalpan
- Moldova (4):
  - Local Institution - 811, Chisinau
  - Local Institution - 809, Chisinau
  - Local Institution - 812, Chisinau
  - Local Institution - 813, Chisinau
- Netherlands (6):
  - Local Institution - 952, Amsterdam
  - Local Institution - 955, Amsterdam
  - Local Institution - 956, Groningen
  - Local Institution - 949, Nijmegen
  - Local Institution - 951, Sittard-Geleen
  - Local Institution - 954, Tilburg
- Poland (56):
  - Local Institution - 403, Zamość, Lublin Voivodeship
  - Local Institution - 597, Zamość, Lublin Voivodeship
  - Local Institution - 820, Bialystok
  - Local Institution - 818, Bochnia
  - Local Institution - 580, Częstochowa
  - Local Institution - 988, Elblag
  - Local Institution - 579, Gdansk
  - Local Institution - 978, Gdansk
  - Local Institution - 577, Gdynia
  - Local Institution - 906, Jelenia Góra
  - Local Institution - 757, Józefów
  - Local Institution - 238, Katowice
  - Local Institution - 578, Katowice
  - Local Institution - 828, Katowice
  - Local Institution - 819, Katowice
  - Local Institution - 815, Krakow
  - Local Institution - 823, Krakow
  - Local Institution - 826, Krakow
  - Local Institution - 834, Ksawerów
  - Local Institution - 817, Kłodzko
  - Local Institution - 581, Lodz
  - Local Institution - 829, Lodz
  - Local Institution - 888, Lodz
  - Local Institution - 981, Lodz
  - Local Institution - 760, Lublin
  - Local Institution - 976, Nowy Targ
  - Local Institution - 830, Olsztyn
  - Local Institution - 402, Opole
  - Local Institution - 400, Oświęcim
  - Local Institution - 758, Poznan
  - Local Institution - 575, Poznan
  - Local Institution - 401, Poznan
  - Local Institution - 963, Rzeszów
  - Local Institution - 979, Sopot
  - Local Institution - 239, Sopot
  - Local Institution - 835, Szczecin
  - Local Institution - 235, Szczecin
  - Local Institution - 822, Torun
  - Local Institution - 824, Tychy
  - Local Institution - 827, Ul. Piotrkowska 177
  - Local Institution - 410, Warsaw
  - Local Institution - 576, Warsaw
  - Local Institution - 833, Warsaw
  - Local Institution - 989, Warsaw
  - Local Institution - 825, Warsaw
  - Local Institution - 236, Warsaw
  - Local Institution - 586, Warsaw
  - Local Institution - 807, Warsaw
  - Local Institution - 893, Wierzchosławice
  - Local Institution - 983, Wroclaw
  - Local Institution - 984, Wroclaw
  - Local Institution - 582, Wroclaw
  - Local Institution - 982, Wroclaw
  - Local Institution - 831, Wroclaw
  - Local Institution - 987, Wroclaw
  - Local Institution - 832, Wroclaw
- Portugal (4):
  - Local Institution - 959, Coimbra
  - Local Institution - 958, Guimarães
  - Local Institution - 961, Loures
  - Local Institution - 957, Viana do Castelo
- Romania (10):
  - Local Institution - 808, Bucharest
  - Local Institution - 836, Bucharest
  - Local Institution - 499, Bucharest
  - Local Institution - 795, Bucharest
  - Local Institution - 837, Bucharest
  - Local Institution - 839, Bucharest
  - Local Institution - 842, Bucharest
  - Local Institution - 838, Cluj-Napoca
  - Local Institution - 843, Craiova
  - Local Institution - 840, Târgu Mureş
- Russia (53):
  - Local Institution - 966, Barnaul
  - Local Institution - 871, Barnaul
  - Local Institution - 589, Bataysk
  - Local Institution - 621, Chelyabinsk
  - Local Institution - 991, Chelyabinsk
  - Local Institution - 598, Chita
  - Local Institution - 848, Irkutsk
  - Local Institution - 882, Kaluga
  - Local Institution - 849, Kemerovo
  - Local Institution - 599, Khanty-Mansiysk
  - Local Institution - 927, Krasnoyarsk
  - Local Institution - 566, Moscow
  - Local Institution - 851, Moscow
  - Local Institution - 873, Moscow
  - Local Institution - 870, Moscow
  - Local Institution - 869, Moscow
  - Local Institution - 990, Nizhny Novgorod
  - Local Institution - 594, Novosibirsk
  - Local Institution - 853, Novosibirsk
  - Local Institution - 876, Novosibirsk
  - Local Institution - 996, Omsk
  - Local Institution - 875, Orenburg
  - Local Institution - 867, Penza
  - Local Institution - 858, Petrozavodsk
  - Local Institution - 859, Pushkin
  - Local Institution - 960, Pyatigorsk
  - Local Institution - 846, Pyatigorsk
  - Local Institution - 883, Rostov-on-Don
  - Local Institution - 863, Saint Petersburg
  - Local Institution - 993, Saint Petersburg
  - Local Institution - 862, Saint Petersburg
  - Local Institution - 868, Saint Petersburg
  - Local Institution - 847, Saint Petersburg
  - Local Institution - 857, Saint Petersburg
  - Local Institution - 845, Saint Petersburg
  - Local Institution - 856, Saint Petersburg
  - Local Institution - 879, Saint Petersburg
  - Local Institution - 878, Saint Petersburg
  - Local Institution - 874, Saint Petersburg
  - Local Institution - 865, Samara
  - Local Institution - 844, Samara
  - Local Institution - 992, Saratov
  - Local Institution - 866, Sochi
  - Local Institution - 806, Tula
  - Local Institution - 881, Ufa
  - Local Institution - 861, Ufa
  - Local Institution - 855, Veliky Novgorod
  - Local Institution - 935, Vladimir
  - Local Institution - 999, Vladivostok
  - Local Institution - 986, Vladivostok
  - Local Institution - 880, Volgograd
  - Local Institution - 583, Yekaterinburg
  - Local Institution - 872, Yekaterinburg
- Saudi Arabia (4):
  - Local Institution - 534, Dammam
  - Local Institution - 537, Jeddah
  - Local Institution - 536, Riyadh
  - Local Institution - 535, Riyadh
- Local Institution - 546, Cape Town, Senegal
- Serbia (12):
  - Local Institution - 241, Belgrade
  - Local Institution - 245, Belgrade
  - Local Institution - 887, Belgrade
  - Local Institution - 246, Belgrade
  - Local Institution - 596, Belgrade
  - Local Institution - 886, Belgrade
  - Local Institution - 890, Belgrade
  - Local Institution - 891, Kragujevac
  - Local Institution - 884, Novi Sad
  - Local Institution - 885, Pančevo
  - Local Institution - 585, Vršac
  - Local Institution - 889, Zrenjanin
- Slovakia (7):
  - Local Institution - 900, Bratislava
  - Local Institution - 894, Bratislava
  - Local Institution - 895, Brezno
  - Local Institution - 899, Nitra
  - Local Institution - 897, Nové Zámky
  - Local Institution - 898, Prešov
  - Local Institution - 896, Rimavská Sobota
- Local Institution - 904, Celje, Slovenia
- South Africa (7):
  - Local Institution - 543, Gauteng
  - Local Institution - 545, Kempton Park
  - Local Institution - 544, Pretoria
  - Local Institution - 542, Pretoria
  - Local Institution - 549, Pretoria
  - Local Institution - 548, Somerset West
  - Local Institution - 547, Val de Grace
- South Korea (15):
  - Local Institution - 437, Ansan
  - Local Institution - 441, Busan
  - Local Institution - 434, Busan
  - Local Institution - 431, Busan
  - Local Institution - 432, Daegu
  - Local Institution - 435, Guri-si
  - Local Institution - 436, Seongnam-si
  - Local Institution - 433, Seoul
  - Local Institution - 440, Seoul
  - Local Institution - 430, Seoul
  - Local Institution - 442, Seoul
  - Local Institution - 438, Seoul
  - Local Institution - 427, Seoul
  - Local Institution - 439, Seoul
  - Local Institution - 429, Suwon
- Spain (16):
  - Local Institution - 703, Alicante
  - Local Institution - 690, Badalona
  - Local Institution - 694, Barcelona
  - Local Institution - 702, Córdoba
  - Local Institution - 699, Girona
  - Local Institution - 701, Las Palmas de Gran Canaria
  - Local Institution - 691, Madrid
  - Local Institution - 695, Madrid
  - Local Institution - 692, Madrid
  - Local Institution - 693, Majadahonda, Madrid
  - Local Institution - 698, San Cristóbal de La Laguna
  - Local Institution - 706, Santander
  - Local Institution - 696, Seville
  - Local Institution - 705, Seville
  - Local Institution - 697, Valencia
  - Local Institution - 700, Viladecans
- Local Institution - 625, Stockholm, Sweden
- Switzerland (3):
  - Local Institution - 967, Bern
  - Local Institution - 968, Sankt Gallen
  - Local Institution - 969, Zurich
- Taiwan (8):
  - Local Institution - 460, Kaohsiung City
  - Local Institution - 463, Kaohsiung, San Ming Dist.
  - Local Institution - 363, Kozlu
  - Local Institution - 461, Niao-Sung Hsiang Kaohsiung County
  - Local Institution - 459, Tainan, Taiana
  - Local Institution - 465, Taipei
  - Local Institution - 462, Taoyuan
  - Local Institution - 464, Tapei, Beitou Dist.
- Turkey (Türkiye) (11):
  - Local Institution - 357, Ankara
  - Local Institution - 356, Ankara
  - Local Institution - 360, Bursa
  - Local Institution - 365, Elâzığ
  - Local Institution - 362, Istanbul
  - Local Institution - 358, Istanbul
  - Local Institution - 361, Istanbul
  - Local Institution - 355, Istanbul
  - Local Institution - 354, Izmit/Kocaeli
  - Local Institution - 353, Kadiköy/Istanbul
  - Local Institution - 359, Trabzon
- Ukraine (38):
  - Local Institution - 914, Chernivtsi
  - Local Institution - 922, Chernivtsi
  - Local Institution - 950, Dnipropetrovsk
  - Local Institution - 229, Ivano-Frankivsk
  - Local Institution - 929, Ivano-Frankivsk
  - Local Institution - 912, Ivano-Frankivsk
  - Local Institution - 919, Kharkiv
  - Local Institution - 965, Kharkiv
  - Local Institution - 920, Khmelnytskyi
  - Local Institution - 933, Kropyvnytskyi
  - Local Institution - 901, Kyiv
  - Local Institution - 923, Kyiv
  - Local Institution - 915, Kyiv
  - Local Institution - 243, Kyiv
  - Local Institution - 563, Kyiv
  - Local Institution - 911, Kyiv
  - Local Institution - 244, Kyiv
  - Local Institution - 564, Kyiv
  - Local Institution - 918, Kyiv
  - Local Institution - 908, Kyiv
  - Local Institution - 977, Kyiv
  - Local Institution - 562, Kyiv
  - Local Institution - 240, Lutsk
  - Local Institution - 590, Lutsk
  - Local Institution - 234, Lviv
  - Local Institution - 974, Lviv
  - Local Institution - 910, Lviv
  - Local Institution - 242, Odesa
  - Local Institution - 902, Odesa
  - Local Institution - 905, Poltava
  - Local Institution - 934, Ternopil
  - Local Institution - 909, Vinnytsia
  - Local Institution - 932, Vinnytsia
  - Local Institution - 224, Vinnytsia
  - Local Institution - 924, Vinnytsia
  - Local Institution - 971, Vinnytsia
  - Local Institution - 587, Zaporizhia
  - Local Institution - 925, Zaporizhzhya
- United Kingdom (15):
  - Local Institution - 723, Southampton, Hampshire
  - Local Institution - 729, London, LND
  - Local Institution - 557, Birmingham
  - Local Institution - 714, Bristol
  - Local Institution - 560, Cardiff
  - Local Institution - 558, Chorley
  - Local Institution - 559, Corbridge Road
  - Local Institution - 712, Dundonald
  - Local Institution - 713, Glasgow
  - Local Institution - 716, Lancashire Blackpool
  - Local Institution - 722, London
  - Local Institution - 715, London
  - Local Institution - 561, North Manchester Science Park
  - Local Institution - 593, Shrewsbury
  - Local Institution - 718, Torquay

REFERENCES:
- [Derived] Feagan BG, Schreiber S, Afzali A, Rieder F, Hyams J, Kollengode K, Pearlman J, Son V, Marta C, Wolf DC, D'Haens GG. Ozanimod as a novel oral small molecule therapy for the treatment of Crohn's disease: The YELLOWSTONE clinical trial program. Contemp Clin Trials. 2022 Nov;122:106958. doi: 10.1016/j.cct.2022.106958. Epub 2022 Oct 5. PMID 36208720
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- RPC01-3201/3202 Placebo; RPC01-3201/3202 Ozanimod 0.92 mg: Responders from the induction study entered the maintenance study. Non-responders had the option to enter the open-label extension 3204 study and took Ozanimod 0.92 mg oral daily.
- RPC01-3203 Placebo-Placebo Completers; RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers; RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers: Participants who completed the 52 weeks maintenance study entered the open-label extension 3204 study and took Ozanimod 0.92 mg oral daily.
- RPC01-3203 Placebo-Placebo Relapse; RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse; RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse: Participants who relapsed in the maintenance study entered the open-label extension 3204 study and took Ozanimod 0.92 mg oral daily.
- RPC01-2201 Ozanimod 0.92 mg: Participants who completed at least 1 year of RPC01-2201 entered the open-label extension 3204 study and took Ozanimod 0.92 mg oral daily.
Period: Overall Study
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg
Started | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13
Not completed — Adverse Event | 20 | 32 | 5 | 3 | 3 | 3 | 6 | 5 | 0
Not completed — Lack of Efficacy | 59 | 120 | 6 | 9 | 8 | 9 | 11 | 9 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Other reasons | 8 | 14 | 2 | 1 | 4 | 0 | 1 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 65 | 117 | 45 | 64 | 66 | 17 | 11 | 5 | 5
Not completed — Withdrawal by Subject | 25 | 44 | 7 | 8 | 6 | 8 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg | Total
Number analyzed (Participants) | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13 | 854
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.93 (13.147) | 39.21 (13.508) | 40.80 (13.988) | 38.21 (13.819) | 41.98 (13.116) | 34.84 (11.100) | 38.06 (12.686) | 39.30 (14.697) | 44.00 (10.368) | 39.10 (13.360)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 151 | 31 | 36 | 48 | 14 | 12 | 11 | 7 | 388
  Male | 101 | 178 | 35 | 49 | 43 | 24 | 21 | 9 | 6 | 466
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 4 | 3 | 4 | 2 | 0 | 0 | 1 | 35
  Not Hispanic or Latino | 168 | 309 | 62 | 81 | 86 | 35 | 29 | 20 | 12 | 802
  Unknown or Not Reported | 3 | 7 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 16 | 35 | 3 | 5 | 5 | 3 | 2 | 1 | 0 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 8
  White | 153 | 274 | 61 | 77 | 82 | 34 | 27 | 19 | 12 | 739
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 17 | 1 | 3 | 2 | 1 | 3 | 0 | 0 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission
Description: Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score of < 150. The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease (CD). The CDAI uses a questionnaire with 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. The sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: At weeks 48, 96, 144, 192, 240
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg
Number analyzed (Participants) | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13
Percentage of participants
  Week 48 | 19.6 | 21.0 | 60.6 | 58.8 | 56.0 | 34.2 | 27.3 | 20.0 | 84.6
  Week 96 | 12.3 | 12.5 | 37.9 | 41.2 | 38.5 | 18.4 | 15.2 | 15.0 | 84.6
  Week 144 | 6.1 | 7.0 | 22.7 | 23.5 | 18.7 | 13.2 | 12.1 | 0 | 61.5
  Week 192 | 4.5 | 4.6 | 6.1 | 11.8 | 9.9 | 2.6 | 3.0 | 5.0 | 30.8
  Week 240 | 2.8 | 3.6 | 1.5 | 3.5 | 1.1 | 2.6 | 0 | 5.0 | 38.5

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) is any AE that emerges or worsens between the day of the first dose of Open-label Extension Study and 90 days after the last dose of Open-label Extension Study. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Serious Adverse Events (SAEs) is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization; results significant disability; or is a congenital anomaly/birth defect.
Time Frame: From first dose to 90 days post last dose (up to approximately an average of 19 months and a maximum of 65 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg
Number analyzed (Participants) | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13
Participants
  TEAE | 140 | 247 | 42 | 63 | 52 | 26 | 22 | 14 | 11
  Serious TEAE | 38 | 59 | 9 | 11 | 11 | 6 | 4 | 2 | 2
  TEAE leading to discontinuation to study drug | 30 | 43 | 4 | 5 | 3 | 4 | 7 | 5 | 1

3. Secondary Outcome: Percentage of Participants With Abdominal Pain (AP) and Stool Frequency (SF) Clinical Remission
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤ 3 points with AP and SF no worse than baseline. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. The AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day. Higher scores indicated worse outcomes.
Time Frame: At weeks 48, 96, 144, 192, 240
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg
Number analyzed (Participants) | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13
Percentage of participants
  Week 48 | 16.2 | 21.3 | 53.0 | 52.9 | 45.1 | 34.2 | 18.2 | 20.0 | 0
  Week 96 | 11.2 | 11.6 | 37.9 | 36.5 | 36.3 | 18.4 | 12.1 | 15.0 | 0
  Week 144 | 5.6 | 7.3 | 21.2 | 24.7 | 14.3 | 13.2 | 12.1 | 0 | 0
  Week 192 | 2.8 | 4.9 | 6.1 | 10.6 | 7.7 | 2.6 | 3.0 | 5.0 | 0
  Week 240 | 3.4 | 3.0 | 1.5 | 1.2 | 1.1 | 0 | 0 | 5.0 | 0

4. Secondary Outcome: Percentage of Participants With Clinical Response
Description: Clinical response is defined as a Crohn's Disease Activity Index (CDAI) reduction from baseline of ≥ 100 points or CDAI score of < 150. The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease (CD). The CDAI uses a questionnaire with 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. The sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: At weeks 48, 96, 144, 192, 240
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg
Number analyzed (Participants) | 179 | 329 | 66 | 85 | 91 | 38 | 33 | 20 | 13
Percentage of participants
  Week 48 | 26.8 | 29.2 | 62.1 | 64.7 | 61.5 | 36.8 | 30.3 | 20.0 | 84.6
  Week 96 | 15.1 | 17.3 | 43.9 | 44.7 | 45.1 | 18.4 | 15.2 | 15.0 | 84.6
  Week 144 | 8.9 | 9.4 | 22.7 | 28.2 | 19.8 | 13.2 | 12.1 | 0 | 61.5
  Week 192 | 5.0 | 6.4 | 6.1 | 12.9 | 11.0 | 2.6 | 3.0 | 5.0 | 30.8
  Week 240 | 3.9 | 4.6 | 1.5 | 3.5 | 2.2 | 2.6 | 0 | 5.0 | 38.5

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 74 months). SAEs and Other AEs were assessed from first dose to 90 days post the last dose (up to approximately an average of 19 months and a maximum of 65 months).
Arm/Group | RPC01-3201/3202 Placebo | RPC01-3201/3202 Ozanimod 0.92 mg | RPC01-3203 Placebo-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers | RPC01-3203 Placebo-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse | RPC01-2201 Ozanimod 0.92 mg
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/329 | 0/66 | 0/85 | 1/91 | 0/38 | 0/33 | 0/20 | 0/13
Serious Adverse Events (participants affected / at risk) | 38/179 | 59/329 | 9/66 | 11/85 | 11/91 | 6/38 | 4/33 | 2/20 | 2/13
Other Adverse Events (participants affected / at risk) | 104/179 | 181/329 | 24/66 | 44/85 | 38/91 | 22/38 | 15/33 | 14/20 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RPC01-3201/3202 Placebo (N=179) | RPC01-3201/3202 Ozanimod 0.92 mg (N=329) | RPC01-3203 Placebo-Placebo Completers (N=66) | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers (N=85) | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers (N=91) | RPC01-3203 Placebo-Placebo Relapse (N=38) | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse (N=33) | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse (N=20) | RPC01-2201 Ozanimod 0.92 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urachal abnormality (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 22 | 24 | 1 | 3 | 2 | 4 | 3 | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal fistula infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leptospirosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RPC01-3201/3202 Placebo (N=179) | RPC01-3201/3202 Ozanimod 0.92 mg (N=329) | RPC01-3203 Placebo-Placebo Completers (N=66) | RPC01-3203 Ozanimod 0.92 Mg-Placebo Completers (N=85) | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Completers (N=91) | RPC01-3203 Placebo-Placebo Relapse (N=38) | RPC01-3203 Ozanimod 0.92 Mg-Placebo Relapse (N=33) | RPC01-3203 Ozanimod 0.92 Mg-Ozanimod 0.92 mg Relapse (N=20) | RPC01-2201 Ozanimod 0.92 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 7 | 17 | 3 | 8 | 4 | 1 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 8 | 1 | 0 | 5 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 13 | 43 | 3 | 7 | 10 | 4 | 3 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Epiretinal membrane (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 18 | 4 | 4 | 2 | 2 | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 4 | 3 | 0 | 1 | 0 | 1 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 33 | 36 | 3 | 7 | 6 | 8 | 4 | 5 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 11 | 2 | 5 | 1 | 0 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 10 | 1 | 3 | 0 | 3 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 11 | 1 | 2 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Medical device pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 11 | 11 | 0 | 4 | 1 | 3 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic dysfunction-associated steatohepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 16 | 25 | 5 | 9 | 15 | 3 | 5 | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 17 | 1 | 4 | 3 | 2 | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 4 | 9 | 0 | 1 | 1 | 2 | 0 | 0 | 2
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 18 | 1 | 0 | 3 | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 9 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood fibrinogen increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 20 | 1 | 2 | 2 | 1 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 1 | 0 | 0 | 1 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 16 | 11 | 3 | 3 | 2 | 3 | 0 | 1 | 0
Morton's neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1 | 2 | 3 | 1 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2 | 1 | 1 | 2 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 5 | 11 | 4 | 1 | 0 | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT03467958/Prot_SAP_000.pdf